CLINICAL TRIAL: NCT04890210
Title: A Comparison of Clear Fluid Diet Initiation Time on Rebleeding Rate and Convenience Level in Liver Cirrhosis Patients Underwent Esophageal Variceal Ligation at Cipto Mangunkusumo Hospital
Brief Title: Initiation of Diet in Esophageal Varices After Ligation (IDEAL) Study
Acronym: IDEAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Rabbinu Rangga Pribadi, MD, Manager of Division of Gastroenterology, Department of Internal Medicine, Dr Cipto Mangunkusumo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DCiptoMGH Indonesia
Record Dates: First submitted 2021-05-06; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Liver Cirrhosis
Keywords: Esophageal Varices After Ligation; Initiation of Diet; Liver cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Diet Group (Experimental): * 1st diet: 100 ml of clear fluid (1 hour after esophageal variceal ligation)
  * 2nd diet: 100 ml of clear fluid (4 hours after the 1st diet)
  * 3rd diet: soft porridge (the amount will be calculated according to patient's caloric needs) which will be given 4 hours after the 2nd diet
  * 4th diet: soft porridge (the amount will be calculated according to patient's caloric needs) which will be given 6 hours after the 3rd diet
  * 5th diet: porridge (the amount will be calculated according to patient's caloric needs) which will be given 6 hours after the 4th diet
  * 6th diet: porridge (the amount will be calculated according to patient's caloric needs) which will be given 6 hours after the 5th diet
  * 7th diet: soft rice (the amount will be calculated according to patient's caloric needs) which will be given 6 hours after the 6th diet
  * 8th diet: regular rice (the amount will be calculated according to patient's caloric needs) which will be given 6 hours after the 7th diet
  Interventions: Dietary Supplement: Early Diet Group
- Late Diet Group (Active Comparator): * 1st diet : 100 ml of clear fluid (6 hours after esophageal variceal ligation)
  * After the 1st diet (Day 1): 6x100 ml of clear fluid for 24 hours
  * Day 2: soft porridge (the amount will be calculated according to patient's caloric needs) for 24 hours
  * Day 3: porridge (the amount will be calculated according to patient's caloric needs) for 24 hours
  * Day 4: soft rice (the amount will be calculated according to patient's caloric needs) for 24 hours
  * Day 5: regular rice (the amount will be calculated according to patient's caloric needs) for 24 hours and beyond
  Interventions: Dietary Supplement: Late Diet Group

INTERVENTIONS:
Dietary Supplement: Early Diet Group — Initiation of clear fluid diet 1 hour after esophageal variceal ligation
  Arms: Early Diet Group
Dietary Supplement: Late Diet Group — Initiation of clear fluid diet 6 hours after esophageal variceal ligation
  Arms: Late Diet Group

SUMMARY:
1. Objective The purpose of this study is to evaluate whether there is a significant difference of early rebleeding rate (within the first 5 days after esophageal variceal ligation), late rebleeding rate (more than 5 days until 28 days after esophageal variceal ligation), and convenience level between cirrhotic patients in early diet group versus late diet group.
2. Method This study is a single blind randomised clinical trial. Subjects will be selected based on inclusion and exclusion criteria, then the subjects will be randomly divided into 2 groups, the early diet group (clear fluid diet is initiated 1 hour after esophageal variceal ligation) and the late diet group (clear fluid diet is initiated 6 hours after esophageal variceal ligation).

   The intervention arm is the early diet group, while the control arm is the late diet group. The primary outcome is the early rebleeding rate. The secondary outcomes are late rebleeding rate and patient's convenience level which will be measured using Visual Analogue Scale (VAS).
3. Expected result The expected result is there will be no difference in early bleeding rate, late bleeding rate, and convenience level between early diet group versus late diet group.

DETAILED DESCRIPTION:
This study is a single blind randomised controlled trial (RCT) that will be conducted at gastrointestinal endoscopy center division of gastroenterology, integrated procedure room division of hepatobiliary, department of internal medicine, gastroenterology clinic, hepatobiliary clinic, internal medicine ward, high care unit (HCU) and intensive care unit (ICU) Cipto Mangunkusumo Hospital - Faculty of Medicine Universitas Indonesia from May 20, 2021-November 1, 2021. The proposed number of subjects are 130 patients.

Interventions will be given in the form of early clear fluid diet initiation compared to active comparator in the form of late clear fluid diet initiation in eligible liver cirrhosis patients who undergo esophageal variceal ligation (EVL) at Cipto Mangunkusumo Hospital. In early diet group diet, the 100 ml of clear fluid will be initiated at 1 hour after EVL followed by standard protocol (clear fluid, soft porridge, porridge, soft rice, regular rice) explained in the arms and intervention column below. In late diet group, the 100 ml of clear fluid will be initiated at 6 hours after EVL, followed by standard protocol (clear fluid, soft porridge, porridge, soft rice, regular rice) explained in the arms and intervention column below. Other routine and standardised drugs for liver cirrhosis patients will still be given. Statistical analysis will use Chi square test with alternative Fisher test for categorical dependent variables and independent T-test with alternative Mann-Whitney test for two group numerical dependent variables.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis patients who underwent esophageal variceal ligation

Exclusion Criteria:

* Hemodynamic instability (shock)
* Possible perforation of the esophagus
* Esophageal diverticula
* Esophageal strictures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-05-20 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Early rebleeding event after esophageal variceal ligation | This outcome (early rebleeding) will be assessed within 5 days after esophageal variceal ligation
  Early rebleeding event is hematemesis, melena and/or hematochezia that occurs within 5 days (120 hours) after esophageal variceal ligation

SECONDARY OUTCOMES:
Late rebleeding event after esophageal variceal ligation | This outcome (late rebleeding) will be assessed between over than 5 days until 28 days after esophageal variceal ligation
  Late rebleeding event is hematemesis, melena and/or hematochezia that occurs between over than 5 days until 28 days after esophageal variceal ligation

OTHER OUTCOMES:
Patient's convenience level regarding initiation of diet after esophageal variceal ligation | Patient's convenience will be measured 30 minutes after the patient finished the 1st clear fluid diet
  Patient's convenience is subjectively measured using Visual Analogue Scale (VAS) 0-10 cm with 0 is very unconvenient and 10 is very convenient

CONTACTS AND LOCATIONS:
Overall Officials: Rabbinu R Pribadi, MD, Principal Investigator — Dr Cipto Mangunkusumo General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Syam AF, Abdullah M, Simadibrata M, Djojoningrat D, Rani A, Manan C. The Causes of Upper Gastrointestinal Bleedingin the National Referral Hospital:Evaluation on Upper Gastrointestinal TractEndoscopic Result in Five Years Period. Indones j gastroenterol. — https://scholar.ui.ac.id/en/publications/the-causes-of-upper-gastrointestinal-bleeding-in-the-national-ref
- See also: Meseeha M, Attia M. Esophageal Varices. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2020 [cited 2020 Jul 8]. — http://www.ncbi.nlm.nih.gov/books/NBK448078/
- See also: Makmun D, Simadibrata M, Fauzi A. Buku Ajar Endoskopi Saluran Cerna. Jakarta: Interna Publishing; 2017. — http://inaactamedica.org/book/book_3.pdf
- See also: Lo G-H, Lin C-W, Hsu Y-C. A controlled trial of early versus delayed feeding following ligation in the control of acute esophageal variceal bleeding. J Chin Med Assoc JCMA. 2015 Nov;78(11):642-7. — http://pubmed.ncbi.nlm.nih.gov/26341455/
- See also: Sidhu SS, Goyal O, Singh S, Kishore H, Chhina RS, Sidhu SS. Early feeding after esophageal variceal band ligation in cirrhotics is safe: Randomized controlled trial. Dig Endosc. 2019 Nov;31(6):646-52. — http://pubmed.ncbi.nlm.nih.gov/31038792/
- See also: Solanki S, Haq K, Chakinala RC,et al. Inpatient burden of esophageal varices in the United States: analysis of trends in demographics, cost of care, and outcomes. Ann Transl Med. 2019 Sep 1;7(18):480. — http://pubmed.ncbi.nlm.nih.gov/31700916/
- See also: Kalista KF, Lesmana CRA, Sulaiman AS, Gani RA, Hasan I. Profil Klinis Pasien Sirosis Hati dengan Varises Esofagus yang Menjalani Ligasi Varises Esofagus di Rumah Sakit Dr. Cipto Mangunkusumo. J Penyakit Dalam Indones. 2019 Mar 31;6(1):36. — http://www.researchgate.net/publication/332150856_Profil_Klinis_Pasien_Sirosis_Hati_dengan_Varises_Esofagus_yang_Menjalani_Ligasi_Varises_Esofagus_di_Rumah_Sakit_Dr_Cipto_Mangunkusumo
- See also: Abby Philips C, Sahney A. Oesophageal and gastric varices: historical aspects, classification and grading: everything in one place. Gastroenterol Rep. 2016 Aug;4(3):186-95 — http://pubmed.ncbi.nlm.nih.gov/27324725/
- See also: . Goda T, Mokhtar A, Anwar R, Hakim H, Eleraki A. Effect of early versus delayed feeding following emergency endoscopic therapy for acute esophageal variceal bleeding on short-term outcomes. Egypt J Intern Med. 2018;30(3):110. — http://ejim.springeropen.com/track/pdf/10.4103/ejim.ejim_22_18.pdf
- See also: Hafeez M. Sucralfate and Lidocain: Antacid 50:50 solution in Post Esophageal Variceal Band Ligation Pain. Pak J Med Sci. 2016 Jul 1;32(4). — http://pubmed.ncbi.nlm.nih.gov/17057145/
- See also: Klimek L, Bergmann K-C, Biedermann T, Bousquet J, Hellings P, Jung K, et al. Visual analogue scales (VAS): Measuring instruments for the documentation of symptoms and therapy monitoring in cases of allergic rhinitis in everyday health care. — http://pubmed.ncbi.nlm.nih.gov/28217433/
- See also: Leigheb M, Sabbatini M, Baldrighi M, et al. Prospective analysis of pain and pain management in an emergency department. — http://pubmed.ncbi.nlm.nih.gov/29083349/